CLINICAL TRIAL: NCT04984772
Title: Understanding Treatment Outcomes of HIV/HBV Coinfection: A Prospective Cohort of HIV/HBV-coinfected Patients in Europe
Brief Title: Prospective Cohort of HIV/HBV-coinfected Patients in Europe
Acronym: Euro-B
Status: Enrolling by invitation | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Euro-B; CO-SW-985-5602 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2021-06-30; First posted 2021-08-02 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections; Hepatitis B; Coinfection
MeSH Terms: conditions — HIV Infections; Hepatitis B; Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma/serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim of the project is to establish an international multi-cohort research platform of HIV/HBV-coinfected individuals treated with tenofovir to improve our understanding of the determinants of treatment outcomes.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is a major cause of morbidity and mortality among human immunodeficiency virus (HIV)-infected individuals and the progression of liver disease is accelerated in this population compared to HBV-monoinfected individuals. Tenofovir disoproxil fumarate (TDF) or tenofovir alafenamide (TAF) as part of antiretroviral therapy (ART) suppresses HBV viral load in most patients. However, risk factors of suboptimal virological response to TDF/TAF and predictors of hepatitis B surface antigen (HBsAg) loss remain unclear. While novel drugs for HBV therapy are being developed, a more thorough understanding of the factors associated with optimal outcomes is urgent. Euro-B considers all HIV/HBV-coinfected participants from EuroSIDA, the Swiss HIV cohort study and French, Spanish and German HIV-HBV cohorts treated with TDF/TAF for inclusion.

The overall aim of the project is to establish an international prospective multi-cohort research platform of HIV/HBV-coinfected individuals to improve our understanding of the determinants of treatment outcomes, including functional cure of HBV infection. Specifically, we aim to:

1. evaluate HBV virological suppression, hepatitis B e antigen (HBeAg) and HBsAg loss as well as the course of quantitative HBsAg (qHBsAg) levels during TDF/TAF-containing antiretroviral therapy
2. evaluate predictors of HBsAg loss and its correlation with Hepatitis B core-related antigen (HBcrAg) and pre-genomic RNA (pgRNA) levels
3. explore risk factors for low-level HBV replication after 2 years of therapy
4. describe changes in liver fibrosis stage and rates of transaminase normalization over time and according to HBV therapy outcome
5. assess rates and reasons of treatment interruptions or changes.

ELIGIBILITY:
Inclusion Criteria:

* Study participant from contributing cohort
* 2 positive HBsAg tests more than 6 months apart
* At least 2 data points (baseline and 2 years after TDF/TAF start either as available data or stored sample

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV/HBV-coinfected individuals treated with tenofovir from Europe
Sampling Method: Non-Probability Sample
Enrollment: 1107 (Estimated)
Dates: Start 2001-10-02 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
HBV suppression | 2 years of TDF/TAF-containing treatment and last available timepoint
  Proportion of participants achieving undetectable HBV DNA
HBsAg loss | 2 years of TDF/TAF-containing treatment and last available timepoint
  Proportion of participants with a negative HBsAg measurement
HBeAg loss | 2 years of TDF/TAF-containing treatment and last available timepoint
  Proportion of participants with a negative HBeAg measurement
Transaminase normalization | 2 years of TDF/TAF-containing treatment and last available timepoint
  Proportion of participants with transaminase normalization
Liver fibrosis change | 2 years of TDF/TAF-containing treatment and last available timepoint
  Proportion of participants with a change in liver fibrosis stage
Treatment interruption or change | 2 years of TDF/TAF-containing treatment and last available timepoint
  Assessments of rates and reasons for treatment interruptions or changes

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Wandeler, MD MSc, Study Chair — Insel Gruppe AG, University Hospital Bern

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Begre L, Boyd A, Plissonnier ML, Testoni B, Beguelin C, Suter-Riniker F, Scholtes C, Rockstroh JK, Lacombe K, Peters L, Heil M, Levrero M, Rauch A, Zoulim F, Wandeler G; Swiss HIV Cohort Study, EuroSIDA and French HIV/HBV and Biliver cohorts; Members of the EuroSIDA Study Group; Members of the French HIV/HBV and Biliver cohorts. Circulating HBV RNA and hepatitis B core-related antigen as determinants of HBsAg loss in persons with HIV in Europe. JHEP Rep. 2025 Nov 7;8(2):101671. doi: 10.1016/j.jhepr.2025.101671. eCollection 2026 Feb. PMID 41551412